CLINICAL TRIAL: NCT07210008
Title: Randomized Controlled Trial Testing the Efficacy of Corticosteroid Therapy Versus Placebo in Fibrotic Hypersensitivity Pneumonitis": RUBY Study (Randomised Trial, glUcocorticoids Versus placeBo in Fibrotic hYpersensitivity Pneumonitis)
Brief Title: "Randomized Controlled Trial Testing the Efficacy of Corticosteroid Therapy Versus Placebo in Fibrotic Hypersensitivity Pneumonitis"
Acronym: RUBY
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP240908; 2025-521591-64-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-22; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Hypersensitivity Pneumonitis
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prednisolone (oral) (Experimental): Prednisolone (oral) will be administered and tapered over 6 months, according to the schedule detailed in the protocol(Cumulative dose: 2430mg/ 6months).
  Active Comparator: prednisolone. Oral prednisolone will be administered and tapered over 6 months, according to the following schedule: 0.5 mg/kg/day (not exceeding 40mg/day) x 4 weeks, 0.25 mg/kg/day (not exceeding 20mg/day) x 4 weeks, 15 mg/day x 4 weeks, 10 mg/days x 4 weeks, 5 mg/day x 10 weeks
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator): Dispersible placebo administered and tapered over 6 months according to the schedule detailed in the protocol
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisolone — Active Comparator: prednisolone. Oral prednisolone will be administered and tapered over 6 months, according to the following schedule*:
  0.5 mg/kg/day (not exceeding 40mg/day) x 4 weeks, 0.25 mg/kg/day (not exceeding 20mg/day) x 4 weeks, 15 mg/day x 4 weeks, 10 mg/days x 4 weeks, 5 mg/day x 10 weeks
  Arms: Prednisolone (oral)
Drug: Placebo — Dispersible placebo administered and tapered over 6 months according to the schedule detailed in the protocol
  Arms: Placebo

SUMMARY:
Hypersensitivity Pneumonitis (HP) is an immune-mediated disease that manifests as interstitial lung disease after exposure to an inhaled antigen, often unidentified. HP can be classified as non-fibrotic or fibrotic HP. Fibrotic HP is associated with impaired quality of life (QoL) and reduced survival. The value and decline of forced vital capacity (FVC) are predictive factors of mortality in fibrotic HP. In most expert centres worldwide, corticosteroids are chosen as the first-line drug to treat fibrotic HP in clinical practice. However, this strategy has not been validated in a randomized controlled trial and it remains controversial, Moreover, corticosteroids are responsible for potentially serious adverse events. The hypothesis is that prednisolone, as a first-line treatment in fibrotic hypersensitivity pneumonitis (HP), slows down FVC decline compared to placebo.

The main objective is to assess the efficacy of first-line treatment with prednisolone against placebo, on the 6-month change in FVC in percent of predicted value (% pred).The primary endpoint will be the absolute change in FVC (% pred) from baseline (inclusion visit,M0) to 6 months (M6) will be compared between the placebo arm and the prednisolone arm.

DETAILED DESCRIPTION:
Hypersensitivity Pneumonitis (HP) is an immune-mediated disease that manifests as interstitial lung disease after exposure to an inhaled antigen, often unidentified. HP can be classified as non-fibrotic or fibrotic HP. Fibrotic HP is associated with impaired quality of life (QoL) and reduced survival. The value and decline of forced vital capacity (FVC) are predictive factors of mortality in fibrotic HP. In most expert centres worldwide, corticosteroids are chosen as the first-line drug to treat fibrotic HP in clinical practice. However, this strategy has not been validated in a randomized controlled trial and it remains controversial, Moreover, corticosteroids are responsible for potentially serious adverse events. The hypothesis is that prednisolone, as a first-line treatment in fibrotic hypersensitivity pneumonitis (HP), slows down FVC decline compared to placebo.

The main objective is to assess the efficacy of first-line treatment with prednisolone against placebo, on the 6-month change in FVC in percent of predicted value (% pred).The primary endpoint will be the absolute change in FVC (% pred) from baseline (inclusion visit,M0) to 6 months (M6) will be compared between the placebo arm and the prednisolone arm.

RUBY, is a national multicenter, randomized, double blind, placebo-controlled, superiority trial comparing the efficacy of prednisolone to placebo on the change in FVC (% pred) at 6 months.

The investigators will randomly assign participants (1:1 ratio, stratification according to the identification of an inciting antigen) to receive oral prednisolone or placebo for a period of 6 months with a follow-up of 12 months. The primary endpoint will be assessed at Month 6.

The investigators plan to include 120 participants.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged above 18 years and under 90 years old
* Diagnosis of fibrotic HP ("definite" or "high confidence") after MDD according to the criteria proposed by guidelines [5]
* Fibrosis extent ≥ 10% on chest HRCT
* Mild to moderate functional impairment defined by FVC ≥ 50% pred and DLco ≥ 30% pred
* Written informed consent for participation in study
* Patient affiliated to a social security scheme or CMU beneficiary
* Effective contraception for men and woman of childbearing age.

Exclusion Criteria:

* Uncertain diagnosis of fibrotic HP ("low confidence" or "unlikely") after MDD according to the criteria proposed by guidelines [5].
* Severe functional impairment defined by FVC < 50% pred and DLco < 30% pred.
* Patient previously treated or currently being treated for fibrotic HP (with corticosteroids, any immunosuppressive agent, or anti- fibrotic therapies).
* Person under guardianship/ curatorship (sous tutelle/curatelle)
* Contraindication to corticosteroid therapy (hypersensitivity to the active substances or to one of the excipients, severe infections, psychotic states not controlled by treatment, live vaccines, uncontrolled diabetes mellitus and uncontrolled arterial hypertension.) or to auxiliary medicinal products
* Patient deprived of liberty under judicial or administrative decision
* Patient participating in another clinical trial with an investigational medicinal product. The patient may participate in another clinical trial after the 6 months of treatment in this study
* Pregnancy or breastfeeding woman
* Patient receiving AME (state medical assistance)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Absolute change in FVC (% pred) | at month 6
  Absolute change in FVC (% pred) from baseline (inclusion visit, M0) to 6 months (M6) will be compared between the placebo arm and the prednisolone arm.

SECONDARY OUTCOMES:
Absolute change in FVC (% pred) according to the presence of a causal antigen at Month 6 | at Month 6
  Absolute change in FVC (% pred) from baseline (M0 or inclusion visit) to Month 6 according to the presence of a causal antigen.
The change in FVC (% pred) at 12 months (M12) | At month 12
  Absolute and relative changes in FVC (% pred) between M0 and M12 will be compared between the placebo arm and the prednisolone arm.
The change in FVC (mL) at 12 months (M12) | At month 12
  Absolute and relative changes in FVC (mL) between M0 and M12 will be compared between the placebo arm and the prednisolone arm.
The changes in DLco (mmol/min/kPa) at Month 6 | At Month 6
The changes in DLco (% pred) at Month 6 | At Month 6
The changes in DLco (mmol/min/kPa) at Month 12 | At Month12
The changes in DLco (% pred) at Month 12 | At Month 12
The changes in distance walked during six-minute walt test 6MWT in meters (m) at Month 12 | at Month12
  Changes in distance walked during 6MWT (m) from Month 0 to Month12 will be compared between the placebo arm and the prednisolone arm
The changes in distance walked during six-minute walt test 6MWT (% pred) at Month 12 | At Month 12
  Changes in distance walked during 6MWT (%pred) from Month 0 to Month12 will be compared between the placebo arm and the prednisolone arm
The changes in distance walked during six-minute walt test 6MWT in meters (m) at Month 6 | At Month 6
  Changes in distance walked during 6MWT (m) from Month 0 to Month 6 will be compared between the placebo arm and the prednisolone arm
The changes in distance walked during six-minute walt test 6MWT (%pred) at Month 6 | At Month 6
  Changes in distance walked during 6MWT (%pred) from Month 0 to Month 6 will be compared between the placebo arm and the prednisolone arm
The change in health related QoL (the Saint Georges Hospital Respiratory Questionnaire (SGRQ) at Month 6 | At Month 6
  Changes in Respiratory QoL (the Saint Georges Hospital Respiratory Questionnaire (SGRQ)) from Month 0 to Month 6 will be compared between the placebo arm and the prednisolone arm
The change in health related QoL (King's Brief ILD questionnaire) at Month 6 | At Month 6
  Changes in Respiratory QoL (King's Brief ILD questionnaire) from Month 0 to Month 6 will be compared between the placebo arm and the prednisolone arm
The change in health related QoL (the Saint Georges Hospital Respiratory Questionnaire (SGRQ) at Month 12 | At Month 12
  Changes in Respiratory QoL (the Saint Georges Hospital Respiratory Questionnaire (SGRQ)) from Month 0 to Month 12 will be compared between the placebo arm and the prednisolone arm
The change in health related QoL (King's Brief ILD questionnaire) at Month 12 | At Month 12
  Changes in Respiratory QoL (King's Brief ILD questionnaire) from Month 0 to Month 12 will be compared between the placebo arm and the prednisolone arm
The proportion of patients who develop pulmonary progressive fibrosis (PPF) within 12 months | Over 12 months
The proportion of subjects who experience acute exacerbation (AE) or require unplanned hospitalization within 12 months | Over 12 months
Progression free survival (PFS) at 12 months | At month 12

CONTACTS AND LOCATIONS:
Overall Officials: Lucile SESE, Study Director — Assistance Publique - Hôpitaux de Paris

IPD SHARING:
Plan to Share IPD: Undecided